CLINICAL TRIAL: NCT03173963
Title: Empagliflozin in Early Diabetic Kidney Disease
Brief Title: Empaglifozin in Early Diabetic Kidney Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Original drug sponsor withdrew from study, replacement sponsor not obtained.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999917103; 17-DK-N103
Record Dates: First submitted 2017-05-27; First posted 2017-06-02 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Diabetic Kidney Disease; Diabetes Mellitus Type 2
Keywords: Sodium Glucose Co-Transporter 2 (SGLT2) Inhibitor; Kidney Biopsy; Morphometry; American Indians; Glomerular Filtration Rate
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug (Active Comparator): Empagliflozin 10mg once a day
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator): 1 placebo tablet a day
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Empagliflozin — 10 mg tablet of empagliflozin daily in addition to best clinical practice for management of diabetes.
  Arms: Drug
Other: Placebo — 1placebo tablet per day
  Arms: Placebo

SUMMARY:
Background:

Diabetes is common among American Indian people and diabetic kidney disease is a common complication. Kidney disease caused by diabetes can lead to the need for kidney replacement, by dialysis or kidney transplant, and is also associated with higher risk of early death. A new diabetes medicine called empagliflozin may slow kidney disease from type 2 diabetes. Researchers want to learn if it protects the kidneys when used in very early stages of diabetic kidney disease.

Objectives:

To see if empaglifozin delays kidney disease development.

Eligibility:

Adults 18-64 years old who are at least half American Indian and have had type 2 diabetes at least 5 years

Design:

Participants will be screened with health questions, blood pressure, and blood and urine tests.

Participants will have:

* Medical history
* Physical exam
* Blood, urine, and stool samples taken
* Scan of the kidneys and liver. Participants will lie on a table that slides into an MRI machine. They will hold their breath for up to 20 seconds and the MRI machine will take images of their kidneys and liver. They will then repeat this with a small device that vibrates on their side.
* Kidney tests. A needle will be placed in a vein in each arm for 4 hours. Blood pressure will be taken. Participants will drink several quarts of water and urinate every 20 minutes. Urine and blood samples will be collected. Two liquids will be injected into their veins to measure kidney function.
* Photos of the back of the eyes
* Kidney biopsy. Participants will have a scan and get drugs to make them sleepy. Up to four very small pieces of kidney will be removed by needle. After the biopsy participants will be monitored for at least 4 hours.
* Nerve tests

Participants will take the study drug or placebo pill once a day. Participants will attend for tests every twelve weeks and have more extensive kidney function tests once a year. After 3 years, participants will have another kidney biopsy and then stop taking the study drug. They will have a final kidney function test 2 months later.

DETAILED DESCRIPTION:
The purpose of this protocol is to examine the effects of the sodium-glucose cotransporter 2 (SGLT2) inhibitor empagliflozin on kidney disease progression in American Indians with type 2 diabetes and early diabetic kidney disease (DKD) via a double-blinded placebo-controlled clinical trial. This trial will enroll 100 participants who will be randomly assigned to receive either 10 mg of empagliflozin or placebo daily for three years in addition to standard of care. Participants will be followed quarterly to monitor their health, identify any adverse effects of treatment, and to assess their adherence to therapy. The primary objective of this study is to determine whether empagliflozin affects structural and functional progression of DKD in American Indians with type 2 diabetes and early DKD to a greater extent than standard diabetes care alone, which may include treatment with renin-angiotensin system (RAS) blockers. The primary outcome measure will be a change in cortical interstitial fractional volume [Vv(Int/cortex)] as assessed by morphometric examination of kidney biopsy specimens obtained at study entry and after the three years of study drug treatment. Secondary outcomes include an effect of empagliflozin on kidney function including measures of glomerular filtration rate and renal plasma flow, and effects on other kidney biopsy morphometric measurements. Biopsy tissue will also be used for gene expression studies and for epigenetic profiling. Magnetic resonance imaging of the kidneys will be performed prior to each biopsy to correlate the structural damage seen at kidney biopsy with the level of fibrosis detected by imaging. In addition to annual renal clearance studies we will conduct a series of other tests at each renal clearance visit. These will include tests of cognitive function and of the peripheral and autonomic nervous system to determine the frequency, severity, and rate of progression of diabetic neuropathy in this cohort and identify linkages between DKD and diabetic neuropathy, and retinal photographs to assess diabetic retinopathy status and its linkage with DKD. The effect of treatment with empagliflozin on the development and progression of neuropathy and retinopathy will also be assessed. To assess acute effects of empagliflozin on renal function at the commencement and cessation of the drug we will undertake additional renal clearance studies two weeks after enrollment and two months after discontinuation of the drug. A small punch skin biopsy may be performed for assessment of intraepidermal nerve fiber density or for fibroblast culture. The skin biopsy for fibroblast culture will be done only once unless the culture fails, in which case the patient may be invited to undergo another biopsy. We may invite participants to undergo skin biopsy on several occassions for assessment of changes in nerve fiber density. We may also perform magnetic resonance imaging of the kidneys or the brain in some participants. Imaging of the kidneys will be done as near to the time of each kidney biopsy as possible. We may invite participants to undergo the brain imaging at the beginning and end of the study. Participants will be followed annually after completion of the clinical trial until death or development of end-stage renal disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for participation in the study, participants must meet the following criteria:

* American Indian heritage participants must be at least half American Indian (i.e. 2 out of 4 grand-parents)
* Aged 18-64 years. The lower age limit was set so renal function test results would not reflect changes associated with growth and the upper limit was set to avoid the bladder emptying problems often encountered in older people, since complete bladder emptying is crucial to the accuracy of the renal function measurements done in this study.
* Diagnosis of type 2 diabetes for greater than or equal to 5 years.
* Estimated GFR >60/ml/min as determined from the CKD-EPI equation using serum creatinine (Levey et al., 2009) or serum creatinine concentration <1.4 mg/dl in women and <1.5 mg/dl in men.
* Serum potassium concentration less than or equal to 5.5 mEq/L.
* A screening urinary albumin-to-creatinine ratio <300 mg/g.
* Willingness to participate after receiving a thorough explanation of the study.
* Participants receiving a RAS blocker must have been receiving the drug for at least 3 months prior to the study baseline examination.

EXCLUSION CRITERIA:

Volunteers will be excluded prior to enrollment for the following reasons:

* Clinically significant disorders of the liver [cirrhosis, portal hypertension, hepatitis, increased bilirubin (greater than or equal to 1.5 mg/dl), cardiovascular disease (angina pectoris, history of myocardial infarction, heart failure, cerebrovascular disease, peripheral vascular disease, pulmonary diseases (asthma and restrictive or obstructive lung disease requiring therapy), renal-urinary disorders (calculi, urinary tract obstruction, glomerulonephritis, chronic infection), gastrointestinal disorders (nausea, vomiting, diarrhea or anorexia sufficient to cause weight loss or wasting), or hematocrit levels less than or equal to 30 percent or >55 percent in women or greater than or equal to 35 percent or >60 percent in men.
* Prior treatment with SGLT2 inhibitors.
* Renovascular or malignant hypertension; uncontrolled hypertension (systolic blood pressure greater than or equal to 160 or diastolic greater than or equal to 95 mm Hg) despite treatment with three antihypertensive drugs.
* Hematuria of unknown etiology. Prior to entry into the study, any participant with hematuria should be evaluated, the etiology established and documented, and treatment rendered as appropriate.
* Chronic debilitating disorders with or without treatment (e.g., systemic lupus erythematosus (SLE), cancer, amyloidosis, and chronic infection) that would interfere with the assessment of kidney function or that might reduce the chances of survival for a sufficient length of time to evaluate the efficacy of treatment.
* Currently receiving a drug regimen that includes: steroids, immunosuppressants, or investigational new drugs.
* Pregnancy. Boerhinger Ingelheim, the manufacturer of empagliflozin, do not recommend its use during the second or third trimester of pregnancy. Moreover, we do not wish to expose pregnant women to conscious sedation that is used during the kidney biopsies or to the intravenous filtration markers iothalamate and para-aminohippurate needed for the renal clearance studies. Women of childbearing potential must have a negative pregnancy test prior to entry and every 3 months during the study, and agree to using an effective form of contraception throughout the study, such as the oral contraceptive pill or an intrauterine device. Women who are planning a pregnancy in the next three years will be excluded.
* Symptoms of inability to empty the bladder. The urinary clearance method is only accurate if complete bladder emptying is possible.
* Hypersensitivity to empagliflozin or iodine.
* Bleeding disorders or requirements for anticoagulation or platelet inhibitors which cannot be safely interrupted, since kidney biopsies cannot be performed safely in these individuals.
* Massive obesity with body mass index greater than or equal to 45 kg/m(2). Kidney biopsies are more difficult and present greater hazards to people with massive obesity.
* Allergy to iodine-containing contrast material.
* Non-diabetic kidney disease based on clinical history or kidney biopsy examination.
* History of severe recurrent kidney infections.
* History of osteoporotic fracture.
* Conditions likely to interfere with informed consent or compliance with the protocol.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-27 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Effect of empagliflozin on change in cortical interstitial fractional volume [Vv(Int/cortex) over the 3-year study period. | 3 years
  Cortical interstitial fractional volume is a measure of the proportion of kidney cortex made up of interstitium. The measurement is made using light microscopy images of kidney tissue. It is positively associated with progression of diabetic kidney disease and is the glomerular measurement that changes most dramatically over time in diabetic kidney disease. We will compare change in cortical interstitial fractional volume from baseline to 3-year biopsy in the group randomized to Empagliflozin and the group randomized to placebo.

SECONDARY OUTCOMES:
Effect of empagliflozin on changes in total interstitium per cortex per kidney, mesangial fractional volume, glomerular basement membrane width, glomerular filtration surface density, and total filtration surface per glomerulus. | 3 years
  Changes in total interstitial volume (calculated from the cortical interstitial fractional volume and cortical volume assessed by MRI) along with key glomerular morphometric measurements (mesangial fractional volume, glomerular basement membrane width, glomerular filtration surface density, and total filtration surface per glomerulus) assessed using electron microscopy images, are all associated with progression of diabetic kidney disease. We will compare change in total cortical interstitial volume and other glomerular measures from baseline to 3-year biopsy in the group randomized to Empagliflozin and the group randomized to placebo.
Effect of empagliflozin on changes in podocyte numerical density, podocyte number per glomerulus, podocyte foot process width, percentage podocyte detachment, and percentage glomerular endothelial cell fenestration. | 3 years
  As diabetic kidney disease progresses podocytes are lost, and the barrier made up of podocyte foot processes and endothelial cell fenestrations becomes more porous. We will compare change in these podocyte measures from baseline to 3-year biopsy in the group randomized to Empagliflozin and the group randomized to placebo.
Effect of empagliflozin on development or progression of diabetic retinopathy determined by changes from baseline to 3 years of at least 2 Early Treatment of Diabetic Retinopathy Study levels in grading of standardized retinal photographs. | 3 years
  Diabetic retinopathy is another microvascular complication of diabetes and untreated can lead to loss of sight. Diabetic retinopathy is detected and staged using digital retinal photography. We will test for effects of Empagliflozin treatment on the incidence of new retinopathy and the progression of existing retinopathy from baseline to 3- years in the group randomized to Empagliflozin and the group randomized to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Looker, Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Cordonnier DJ, Pinel N, Barro C, Maynard M, Zaoui P, Halimi S, Hurault de Ligny B, Reznic Y, Simon D, Bilous RW. Expansion of cortical interstitium is limited by converting enzyme inhibition in type 2 diabetic patients with glomerulosclerosis. The Diabiopsies Group. J Am Soc Nephrol. 1999 Jun;10(6):1253-63. doi: 10.1681/ASN.V1061253. PMID 10361863